CLINICAL TRIAL: NCT02884986
Title: Randomised Controlled Trial - Multimodal Analgesia in Inguinal Hernia Repair Using a Cyclooxygenase-2-specific Inhibitor: A Randomised Controlled Trial
Brief Title: Analgesia in Inguinal Hernia Repair Using a Cyclooxygenase-2-specific Inhibitor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS.GAITINI, M.D., Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BnaiZionMC-16-LG-009
Record Dates: First submitted 2016-08-17; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Adverse Anesthesia Outcome
Keywords: Etoricoxib; Spinal anaesthesia; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etoricoxib (Active Comparator): 120mg of oral Etoricoxib under the brand name Arcoxia® (Merck Sharp & Dohme) one hour prior to spinal anaesthesia induction
  Interventions: Drug: Etoricoxib
- Placebo (Placebo Comparator): 120mg of oral Placebo the same amount as the drug administrated one hour prior to spinal anaesthesia induction
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etoricoxib — 120mg of oral etoricoxib under the brand name Arcoxia® (Merck Sharp & Dohme) one hour prior to spinal anaesthesia induction
  Arms: Etoricoxib
Drug: Placebo — 120mg of placebo
  Arms: Placebo

SUMMARY:
Acute pain is the result of activating nociceptive pathways in both the peripheral and central nervous system. The origin of most acute pain from surgical stimulation is the mechanical trauma of the local tissue and the subsequent acute inflammatory response.

No studies have investigated the combined use of anti-inflammatory analgesics with spinal anaesthesia/analgesia for pre, intra and postoperative multimodal pain protection in patients undergoing day-case IHR. The aim of the investigators study is therefore to assess the efficacy of preoperative combined administration of etoricoxib and standard spinal anaesthesia in the reduction of postoperative pain following IHR.

DETAILED DESCRIPTION:
Acute pain is the result of activating nociceptive pathways in both the peripheral and central nervous system. The origin of most acute pain from surgical stimulation is the mechanical trauma of the local tissue and the subsequent acute inflammatory response. Open inguinal hernia repair is one of the commonest surgical procedures which may provoke pain of variable intensity and duration.

Etoricoxib (Arcoxia®) is a NSAID with anti-inflammatory and analgesic properties mainly achieved via selective peripheral COX-2 inhibition. Spinal anaesthesia using local anaesthetics combined with opioids affects the transmission, modulation and modification stages of nociceptive afferent impulses and its analgesic qualities are superior to local anaesthesia alone.

No studies have investigated the combined use of anti-inflammatory analgesics with spinal anaesthesia/analgesia for pre, intra and postoperative multimodal pain protection in patients undergoing day-case IHR. The aim of the investigators study is therefore to assess the efficacy of preoperative combined administration of etoricoxib and standard spinal anaesthesia in the reduction of postoperative pain following IHR.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiology Class I and II

Exclusion Criteria:

* Under treatment with Non Steroid Antinflammatory Drug
* Under Opioid treatment
* Peptic ulcer
* Liver insufficiency
* Renal insufficiency
* Asthma
* Cardiovascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pain VAS Score | Each four hours until 24 hours
  In the post operative period

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Gaitini, M.D., Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes